CLINICAL TRIAL: NCT01402453
Title: Monetary Incentives and Intrinsic Motivation to Sustain Hypertension Control Pilot Study
Brief Title: Monetary Incentives and Intrinsic Motivation to Sustain Hypertension Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Martin Shapiro, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 11-008320; 1RC4AG039077-01 (NIH)
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension
Keywords: Incentives; Social psychology; Randomized trial; Hypertension; Intervention; Pilot Study
MeSH Terms: conditions — Hypertension | interventions — Economics, Behavioral; Psychology, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Subjects (No Intervention): Receive educational materials and a home BP monitor.
- Intervention Subjects (Experimental): Receive educational materials and a home BP monitor, as well as monetary incentives tied to amount of improvement in BP from baseline and a personalized intervention to internalize motivation for BP control. Monthly monetary incentives will cease after 6 months.
  Interventions: Behavioral: Monetary Incentives; Behavioral: Intrinsic Motivation

INTERVENTIONS:
Behavioral: Monetary Incentives — Subjects will receive a payment of $2 per mm. drop in BP from the baseline value at each follow-up visit. If a subject reaches their target BP, they will receive a minimum of $30 each time to motivate continued participation in the study and reinforce continued improvement relative to baseline BP. Lottery incentives will be added to motivate attainment of intermediate goals. For remembering to do certain actions that assist in the management of their BP, the subject will receive one entry into a lottery with an expected value of $3 per ticket. For the lottery payment, the subject will be given 3 chances to randomly select a card that may or may not show a winning monetary prize.
  Other Names: Behavioral economics
  Arms: Intervention Subjects
Behavioral: Intrinsic Motivation — A)Subjects will complete an additional component to the baseline questionnaire that probes systematically for areas of experience that currently are of importance to them. Their answers will help to identify patients' intrinsic motivations for controlling their BP. B)Answers to this component will be analyzed to characterize a role self-identity that will be used by study personnel to frame their interactions with the subject for the remainder of the study. C) Role identity will be kept highly salient throughout the study by using identity primes that remind the individual that improving blood pressure levels is an important responsibility associated with that role.
  Other Names: Social Psychology
  Arms: Intervention Subjects

SUMMARY:
Despite unequivocal proof that tight control of blood pressure with antihypertensive medication can prevent hypertensive complications-including strokes, myocardial infarcts, heart failure, end-stage renal disease, and death- blood pressure remains uncontrolled in the majority of individuals with hypertension. We propose a novel patient-centered intervention that combines monetary incentives and a social psychological intervention to help patients sustain blood pressure control once incentives are no longer offered by strengthening intrinsic motivation to control blood pressure among two vulnerable populations: African Americans, who suffer disproportionately from hypertension, and Mexican Americans, who have the lowest hypertension control rates of any demographic group in the United States. If the intervention is successful, it could be adapted as a set of tools to apply in clinical practice to improve outcomes of a range of chronic diseases, by maximizing the motivation of patients to optimize their treatment.

DETAILED DESCRIPTION:
We propose to test the translation of behavioral economics and social psychology theory and experience in other domains into an intervention that has the potential to improve control of hypertension and diminish its health impact. Blood pressure control requires that: (1) the patient see a physician; (2) the disease be recognized by the physician, (3) a medicine be prescribed; (4) the patient take the medicine; (5) the patient come back for additional visits to monitor the treatment; (6) the provider make adjustments as needed in the therapy; and (7) the patient adhere to the changes and continue to come in for monitoring. Factors interfere with this chain of events even among patients with a regular source of care, such as a community clinic. Due to the asymptomatic nature of the disease, lack of awareness of the consequences of uncontrolled BP, discounting of these consequences because they occur in the distant future, health beliefs that lead the individual not to believe that the treatment would be beneficial, competing demands, financial barriers, or medication side effects, these patients may not monitor their BP as often as they should, press their physicians about BP control, or adhere to medication regimens. For their part, physicians may not intensify treatment as indicated.

How would the combination of incentives that we propose in this study work in hypertension management? Monetary incentives could improve BP control by leading patients to monitor their BP and make physician visits for hypertension more frequently, "activating" patients to be more assertive about discussing treatment intensification with their providers when their BP is elevated or other issues regarding their therapy, and improving medication adherence. Thus a patient whose BP readings continue to be elevated because he or she is receiving inadequate monotherapy for their level of hypertension might be more motivated to remember to take their pills, check their readings regularly, and most importantly, get to the doctor to intensify the regimen when faced with a monetary incentive to reduce BP. Similarly, another patient might be more motivated to speak up and tell their physician that they are having trouble taking their current BP medicine because of its side-effects; rather that stopping their medication and suffering the consequences of uncontrolled hypertension, this "activated" patient may stimulate the physician to prescribe a different class of medicine that effectively controls the BP without side-effects. Although this experience may give the patient insight that they can get their blood pressure under control and keep it there for some time, the same concerns that initially interfered with BP control may lead patients to return to previous habits after the monetary incentive is withdrawn. They may be busy and not make the time to check their blood pressure, refill prescriptions, take their medicine, or see their doctor. For this reason, helping the patient identify intrinsic motivations to control their BP is necessary. Intrinsic motivations would help keep the patient continually aware of what is at stake (in terms of the people they care about, their roles in society, and their activities) if they do not take their medicines, fill their prescriptions, or follow up with the provider when blood pressure readings are not at target.

The challenge of achieving and sustaining hypertension control might usefully borrow terminology from clinical oncology, in which many treatments have 3 phases: induction, consolidation, and maintenance. For hypertension, we can envision a similar framework: induction of normal blood pressure through initiation and adjustment of medications and adherence to them (for which we expect monetary incentives to be most effective); consolidation in which the patient maintains a normal blood pressure for a period of time (reinforced by frequent feedback, ongoing incentives, and interventions aimed at making intrinsic motivations salient); and maintenance after withdrawal of the incentives, which can be reinforced by success reducing blood pressure coupled with identity priming and identity labeling to engender strong intrinsic motivation to continue.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or older who are receiving ongoing medical care at the clinic (one or more routine visits in the year prior to the visit during the study enrollment period at which their blood pressure is found to be abnormal), are capable of giving consent, and live at a fixed address.
* Must state that they intend to continue to receive care in the clinic.
* Measured BP is greater than 140mm systolic or 90mm diastolic (or 130/80 respectively for "high risk" subjects with: diabetes, established coronary artery disease, prior cardiovascular event, left ventricular hypertrophy by ECG, chronic kidney disease, or diagnosed heart failure).

Exclusion Criteria:

* Those whose BP's have returned to normal 1-2 weeks after the original obtained average reading.
* Children, prisoners, institutionalized individuals, or pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in and normalization of BP | 12 months

SECONDARY OUTCOMES:
Acceptability of the intervention and subjects' views regarding its impact. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin F. Shapiro, MD, Principal Investigator — University of California, Los Angeles; José J. Escarce, MD, Ph.D, Study Director — University of California, Los Angeles; Craig R. Fox, Ph.D., Study Director — University of California, Los Angeles; Noah J. Goldstein, Ph.D., Study Director — University of California, Los Angeles; Honghu Liu, Ph.D., Study Director — University of California, Los Angeles; Suzanne B. Shu, Ph.D., MBA, Study Director — University of California, Los Angeles; Ronald G. Victor, MD, Study Director — Cedars-Sinai Medical Center for Hypertension
Locations (2):
- United States (2):
  - St. John's Well Child and Family Center Compton W.M. Keck Foundation Clinic Building, Los Angeles, California
  - St. John's Well Child and Family Center Dr. Louis C. Frayser Clinic, Los Angeles, California

REFERENCES:
- [Derived] Shapiro MF, Shu SB, Goldstein NJ, Victor RG, Fox CR, Tseng CH, Vangala S, Mogler BK, Reed SB, Villa E, Escarce JJ. Impact of a Patient-Centered Behavioral Economics Intervention on Hypertension Control in a Highly Disadvantaged Population: a Randomized Trial. J Gen Intern Med. 2020 Jan;35(1):70-78. doi: 10.1007/s11606-019-05269-z. Epub 2019 Sep 12. PMID 31515735